CLINICAL TRIAL: NCT01722461
Title: A Prospective, Multi-Center, Parallel, Randomized, Double-Blinded Study of the Efficacy and Safety of the Ulthera® System for the Treatment of Primary Axillary Hyperhidrosis
Brief Title: A Study of the Ulthera® System for the Treatment of Axillary Hyperhidrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision; unexpectedly high sham response at primary outcome time point.
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ULT-119
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-12

CONDITIONS: Primary Axillary Hyperhidrosis
Keywords: Excessive underarm sweating

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active treatment (Experimental): Ulthera System treatment
  Interventions: Device: Ulthera System
- Sham treatment (Sham Comparator): Ulthera System delivering no ultrasound energy
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: Ulthera System — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™
  Arms: Active treatment
Device: Sham treatment — Ulthera System delivering no ultrasound energy
  Arms: Sham treatment

SUMMARY:
This is a prospective, multi-center, randomized, double-blinded study. Subjects enrolled will be randomly assigned to receive either active treatments for axillary hyperhidrosis with the Ulthera System in both axillas, or sham treatments, also with the Ulthera System but with the energy settings on the device set to deliver no ultrasound energy. Subjects will be randomized in a 2:1 ratio, with 2 subjects randomized to active treatment for every one subject randomized to sham treatment. Subjects will receive 2 study treatments 30 days apart.

Subjects and study personnel conducting efficacy measures will be blinded to the assigned treatment groups. The study hypothesis is that subjects in the active treatment group will have a greater reduction in underarm sweating compared to those in the sham group as measured by a quality of life questionnaire.

All subjects will undergo follow-up assessments at 14 days and 30 days from the date of their first study treatment, and 14 days, 30 days, 3 months and 6 months from the date of their second study treatment. Subjects in the active treatment group will also undergo follow-up assessments at 9 months and 12 months from the date of their second study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, age 18 years or older.
* Subject is in good health.
* Diagnosis of primary focal axillary hyperhidrosis evidenced by at least two of the standard criteria.
* At least 50mg at 5 min of spontaneous resting axillary sweat production in each axilla measured gravimetrically
* A HDSS score of 3 or 4
* Willingness to comply with study visits and requirements
* Female subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at Visit 1
* Female subjects over 40 years of age must have had a mammogram in the last 2 years

Exclusion Criteria:

* Has a dermal disorder including infection at anticipated treatment sites in either axilla.
* Has had axillary injections of botulinum toxin in the last year.
* Has an expected use of botulinum toxin for the treatment of any other disease during the study period.
* Has a known allergy to starch powder, iodine, or lidocaine.
* Has secondary hyperhidrosis
* Has had previous surgical treatment of hyperhidrosis
* Has had prior miraDry treatment for axillary hyperhidrosis.
* Has used prescription antiperspirants in the last 14 days or plans to use them during the study period.
* Inability to withhold use of non-study-supplied antiperspirants and deodorants
* Unwillingness to wash off study-supplied antiperspirants and abstain from use for 72 hours prior to treatments or assessments.
* History of previous Ultherapy™ treatment to the axilla.
* Has a history of a bleeding disorder
* Has used of cholinomimetics, anticholinergics, or any oral herbal medicine treatments for hyperhidrosis in the past 4 weeks.
* Is a prisoner or under incarceration.
* Is participating in another clinical trial involving the use of investigational devices or drugs (or has in the last 30 days.)
* Has a history of cancer (some exceptions), lymphectomy, or a planned lymphectomy.
* Has a pacemaker or other electronic implant.
* Requires supplemental oxygen.
* Has used antiplatelet agents / Anticoagulants (Coumadin, Pradaxa, Heparin, Plavix) in the past 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Percentage of active treated subjects compared to sham treated subjects with reduced underarm sweating | 30 days post-treatment #2
  As measured by the Hyperhidrosis Disease Severity Scale (HDSS), a quality of life questionnaire

SECONDARY OUTCOMES:
Percentage of active treated subjects compared to sham treated subjects with reduced underarm sweating | 6 month post treatment #2
  As measured by the HDSS
Percentage of active treated subjects compared to sham treated subjects with reduced underarm sweating | 12 months post treatment #2
  As measured by the HDSS
Percentage of active treated subjects compared to sham treated subjects with reduced average spontaneous axillary sweat production | 3 months post treatment
  As measured by gravimetric method
Percentage of active treated subjects compared to sham treated subjects with reduced spontaneous axillary sweat production | Subjects will be followed to 12 months post treatment #2
  As measured by gravimetric method

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nestor, M.D., Ph.D, Principal Investigator — The Center for Clinical and Cosmetic Research
Locations (6):
- United States (6):
  - Roseville Facial Plastic Surgery, Roseville, California
  - The Center for Clinical and Cosmetic Research, Aventura, Florida
  - Few Institute of Aesthetic Plastic Surgery, Chicago, Illinois
  - St Louis University Dermatology, St Louis, Missouri
  - Day Dermatology & Aesthetics, New York, New York
  - Virginia Clinical Research, Norfolk, Virginia